CLINICAL TRIAL: NCT04699006
Title: The Efficacy and Adverse Effects of Olaparib in Ovarian Cancer: a Prospective Real-world Product Registration Study.
Brief Title: Efficacy and Adverse Effects of Olaparib in Ovarian Cancer.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2020LSK-205
Record Dates: First submitted 2020-12-17; First posted 2021-01-07 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-12

CONDITIONS: Ovarian Cancer
Keywords: olaparib; real word; prospective; efficacy and adverse effects; product registration study
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20ml blood samples and surgically removed histological samples of enrolled patients are collected (only for enrolled patients who agree to blood sampling) for exploratory biological marker research and exploratory pharmacogenetic analysis. All collected specimens will be kept in the first affiliated Hospital of Xi'an Jiaotong University.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ovarian cancer is the second fatal gynecological cancer. More than 70% of ovarian cancer patients are diagnosed as advanced. Olaparib is the first oral poly adenosine diphosphate-ribose polymerase inhibitor (PAPPi) approved by the U.S. Drug Administration (FDA) in December 2014. It can be used as a maintenance treatment for adult patients with platinum-sensitive recurrent epithelial ovarian cancer, fallopian tube cancer, and primary peritoneal cancer after platinum-containing chemotherapy has achieved complete or partial remission. At present, most studies based on olaparib are randomized controlled trials (RCTs). Because RCTs often have strict inclusion and exclusion criteria and they are implemented in a highly standardized environment. Its internal validity is high, but the research results may not be able to be extrapolated to practice. This study is a prospective real world study. In this study, based on the modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1), we evaluate the use of olaparib in patients with ovarian cancer, fallopian tube cancer, and primary peritoneal cancer in the progression-free survival (PFS), overall survival (OS), and objective control rate (ORR), etc. At the same time, the safety and tolerability of olaparib and the impact on the quality of life of patients are evaluated. Finally, we analyze the results as a supplement to the conclusions of randomized controlled trials to provide better guidance for patients.

DETAILED DESCRIPTION:
1. Research status at domestic and foreign

   Ovarian cancer is the second fatal gynecological cancer. More than 70% of ovarian cancer patients are diagnosed as advanced. Standard treatments include optimal reduction surgery and platinum/taxane chemotherapy. Epithelial ovarian cancer (EOC) is the most common histological type of ovarian cancer, up to 20% of high-grade serous ovarian cancer (HGSOC) shows germline and/or somatic mutations in the BRCA1/BRCA2 gene. BRCA1 and BRCA2 are tumor suppressor genes that play a central role in repairing DNA double-strand breaks (DSBS) through homologous recombination (HR). Due to their increased sensitivity to DNA damage reagents, they extend the survival period of BRCA1 and BRCA2 mutant EOCs, among which BRCA2 vectors have the best survival rate. Poly-adenosine diphosphate-ribose polymerase 1 is a key ribozyme involved in single-strand break (SSB) repair through the base excision repair pathway. In the absence of poly adenosine diphosphate-ribose polymerase(PARP) activity, these lesions are considered to have transformed into DSB. Cells lacking HR, such as BRCA mutant cells, are extremely sensitive to PARP inhibition. This phenomenon called "synthetic lethality" has led people to study poly adenosine diphosphate-ribose polymerase inhibitors (PARPi) used as therapeutic agents in BRCA1/BRCA2 carriers.

   Olaparib is the first oral PARPi approved in the United States in December 2014 for the fourth-line treatment of advanced ovarian cancer with BRCA mutations. In the early development of PARPi olaparib, studies have found that platinum sensitivity seems to be related to a higher objective response rate between BRCA carriers and non-carriers. Gelmon et al. designed a phase II randomized trial Study 19, which evaluated the efficacy of olaparib and placebo as maintenance therapy in patients with platinum-sensitive serous ovarian cancer recurrence. Compared with the placebo group, the median progression-free survival (PFS) of the olaparib group was significantly longer (8.4 months for the olaparib group and 4.8 months for the placebo group (HR=0.35; [95) % credibility interval (CI) =0.25-0.49]; p<0.001). Post-hoc analysis showed that among BRCA germline mutations (gBRCA) carriers, the improvement of PFS in the olaparib group was greater (HR≤0.18; [95%CI=0.10-0.31]; p <0.0001). The SOLO2 study is a randomized, controlled phase III randomized controlled trial, which further confirmed the findings of patients with gBRCA mutations in Study 19. At present, based on the latest National Comprehensive Cancer Network (NCCN) guidelines and guidelines for the clinical application of PAPPi for ovarian cancer, the first-line recommends PARPi+bevacizumab (Bev) maintenance therapy, and PARPi maintenance therapy is the standard treatment for platinum-sensitive recurrent epithelial ovarian cancer.

   The above-mentioned studies based on olaparib are mostly randomized controlled trials (RCTs). Because RCTs often have strict inclusion and exclusion criteria, they are carried out in a highly standardized environment, so that the research subjects have good homogeneity. The validity is high, but the research results may not be able to be extrapolated to practice. Therefore, it is necessary to evaluate the role of treatments for advanced diseases in the real world. To provide better guidance for patients, real-world evidence is needed to make up for the lack of randomized controlled trials. At present, in real-world researches, there are only retrospective studies on the use of olaparib in ovarian cancer at home and abroad, and the results are consistent with its corresponding RCTs. There is a lack of prospective real-world evidence with higher levels of evidence.
2. Study drugs

   The drug name is olaparib tablets. This product is a film-coated tablet. 1)150mg: green to green/gray, oval, biconvex tablets, with "OP150" engraved on one side and blank on the other side. 2)100mg: yellow to dark yellow, oval, biconvex tablets, with "OP100" engraved on one side and blank on the other side.
3. Research programs

   3.1 Overall design

   This study is a prospective real-world product registration study. It is an observational study. The main research content is to evaluate the efficacy and adverse reactions of PARPi olaparib in patients with ovarian cancer, fallopian tube cancer or primary peritoneal cancer. According to the inclusion and exclusion criteria, we collect various information of the target research participants, and organize the data and perform statistical analysis under the guidance of epidemiologists and statistical experts. The curative effect is evaluated by indicators such as PFS, overall survival (OS), and objective response rate (ORR). Moreover, we collect and analyze the adverse reactions of study participants after taking olaparib. 20ml blood samples and surgically removed histological samples of enrolled patients are collected (only for enrolled patients who agree to blood sampling) for exploratory biological marker research and exploratory pharmacogenetic analysis.

   3.2 Sample size

   This research is an observational study. 245 study participants are expected to be included.

   3.3 Stratification factors

   This research can set up different plans according to the following different stratification factors and research purposes.1) Number of treatment lines: first-line maintenance, second-line maintenance, back-line treatment, excess indications. 2) BRCA1/2 mutation status: positive, negative. 3) Platinum sensitive status: platinum sensitive, platinum resistant. 4) CA125 level, etc.

   3.4 Treatment plan

   This study is a non-interventional study that only collects data and does not interfere with clinical treatment. The medication is administered according to clinical instructions, guidelines and local treatment routines.
4. Research process

   4.1 Subject informed

   Patients should sign an informed consent form before the start of the study. The researchers need to explain the contents of the informed consent to the subjects in detail. After the candidate has fully read and understood the informed consent, if she agrees to participate in the study, the subject should sign and date the informed consent. Researchers also need to sign and date the informed consent form.

   4.2 Interview on selection

   Within 7 days of the subjects' enrollment, the investigator collected baseline data, including: general information; medical history diagnosis; past tumor treatment history; family history; whether it meets the admission criteria.

   4.3 Interview during treatment and the last interview

   After the subjects are enrolled, the investigator will conduct a visit every 12 weeks. The data include:
   * Efficacy evaluation: CT/MRI imaging examination and tumor marker CA125 examination are required.
   * Safety evaluation: whether there are adverse events (AE).
   * At baseline, at the same time as the RECIST assessment time (once every 12 weeks) until the objective radiation disease progression or the end of the study treatment interview, a functional assessment of cancer treatment-ovarian cancer (FACT-O) questionnaire survey.
5. Safety evaluation

   5.1 Definition of Adverse Events

   AE refers to all the adverse medical events that occur after the subject receives the experimental drug. It can be manifested as symptoms and signs, diseases or abnormal laboratory tests, but it may not be causally related to the experimental drug.

   5.2 Severity of adverse events

   During the study period, the severity of AEs will be classified according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0, and AE of grade ≥3 will be collected.

   5.3 Relationship with study drug

   When judging the correlation between AEs and study drugs, the following factors should be considered: 1) It is definitely related; 2) It may be related; 3) Possibly irrelevant; 4) Definitely irrelevant; 5) Undecidable.

   5.4 Adverse event records

   All adverse events that occur from the subject's first use of olaparib to 4 weeks after the last dose, including observed by the investigator, obtained by inquiries, and spontaneously reported by the subject should be fully recorded.

   Researchers need to continue to follow up all AEs until the event is cured, returns to baseline, reaches a stable state, or no more information is available. The researcher needs to monitor and record the outcome of the AE in the subject's source file. After the study, there is no need to actively collect new AEs.
6. Drug management

   This study is a real-world study, and olaparib is a marketed drug, so olaparib needs to be purchased and used by patients according to the normal procedures in the hospital.
7. Data recording and monitoring

   7.1 Data logging

   This project uses table records. According to Good Clinical Practice (GCP) requirements, in order to ensure patient privacy, patient names should not appear. All patients' names should be filled with name codes, and the codes should be abbreviated in Chinese name. The specific dosage and time of medication are unknown, and should be filled in unknown rather than blank or missing items. The researcher should ensure that all data must be consistent with the "inpatient medical record".

   7.2 Data monitoring

   During the test process, the research unit will review the completed test case data, check whether the data is correct, complete and standardized, and assess the traceability of all data.
8. Statistical analysis

   8.1 Definition of statistical analysis data sets

   The study includes cases that have received at least one trial drug and have a safety evaluation into the primary and secondary endpoint analysis. Those who have not used a trial drug or have no research data after being selected can be eliminated. Excluded cases should be kept for future reference and no statistical analysis should be performed.

   8.2 Statistical analysis methods

   The continuous variables in this study are described by median and interquartile range. Categorical variables are described by absolute value and the proportion of the total number of patients. Χ2 test are used for comparison between groups. The method of survival analysis is used to statistically process the follow-up data. Kaplan-Meier method is used to draw the survival curve of the follow-up subjects. Log-Rank test was used to evaluate the survival difference between each group. Cox regression model was used to analyze the influencing factors of the survival time of each group of follow-up subjects. Candidate influencing factors with a significance level of 0.05 in the univariate analysis were selected into the multivariate analysis. For all analyses, the test level α=0.05, when p<0.05 is considered statistically significant. All analyses were performed using Statistical Product and Service Solutions (SPSS) software (version 22.0).
9. Quality control and quality assurance

All research processes should establish standardized operating procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary ovarian cancer, fallopian tube cancer, or peritoneal cancer confirmed by histology.
2. Patients who are taking olaparib.
3. Patients should voluntarily participate in the trial and provide signed informed consent.

Exclusion Criteria:

1) Patients who are not currently taking olaparib treatment.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are taking olaparib who suffer from primary ovarian cancer, fallopian tube cancer, or peritoneal cancer confirmed by histology.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  PFS is defined as the time from the first day of olaparib administration to disease progression (defined as objective radiological disease progression using modified Recist version 1.1 or clinical progression) or death.
Adverse event(AE) | 24 months
  Adverse Event (AE) refers to all the adverse medical events that occur after the subject receives the experimental drug. It can be manifested as symptoms and signs, diseases or abnormal laboratory tests, but it may not be causally related to the experimental drug.

SECONDARY OUTCOMES:
Overall survival (OS) | 60 months
  OS is defined as from the first day of administration of olaparib to death of any cause or the patient's last follow-up.
Objective response rate (ORR) | 24 months
  ORR refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including complete response (CR) + partial response (PR) cases. CR refers to the disappearance of all target lesions, including normal tumor markers and no new lesions at least 4 weeks. PR refers to a reduction in the sum of the maximum diameter of the target lesion by ≥30%, which is maintained for at least 4 weeks.
Health-related quality of life (HRQoL) | 24 months
  The functional assessment of cancer treatment-ovarian cancer (FACT-O) test result index (TOI) is used to assess the health-related quality of life of patients reported.

OTHER OUTCOMES:
BRCA1/2 mutation status | 24 months
  The BRCA1/2 mutation status of the tumor.
Platinum sensitivity status | 24 months
  The correlation between platinum sensitivity status and efficacy.
Histological classification | 24 months
  The correlation between histological classification and efficacy.
CA-125 level | 24 months
  The correlation between CA-125 level and efficacy.
Retrospective biomarker & genetic pharmacology studies (optional). | 24 months
  Possible retrospective biomarker & genetic pharmacology studies (optional) are evaluated in accordance with clinical routine cycles and requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Qiling Li, MD,PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China